CLINICAL TRIAL: NCT03876964
Title: J-Valve Compassionate Use Cases
Brief Title: J-Valve Compassionate Use
Status: No longer available | Type: Expanded Access
Sponsor: JC Medical, Inc., an affiliate of Edwards Lifesciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: JCU-001
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Disease; Aortic Valve Insufficiency; Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Insufficiency; Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Device: Transcatheter Aortic Valve Replacement — Minimally invasive replacement of the aortic valve through a catheter.
  Other Names: TAVR

SUMMARY:
J-Valve TF Compassionate Use cases approved on a case by case basis by the FDA

DETAILED DESCRIPTION:
The J-Valve is designed to treat patients with aortic valve disease requiring replacement. There are certain patient subsets that the J-Valve TF is uniquely able to treat and where there are no good alternative treatments for patients at high surgical risk. Physicians have applied for individual approval to treat patients with the J-Valve in certain clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult